CLINICAL TRIAL: NCT03647137
Title: Amyloidopathy, Cholinopathy, Dopamine Responsiveness and Freezing of Gait in PD
Acronym: FOG
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: B1631-I; HUM00110351 (Other: University of Michigan)
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Parkinson's Disease
Keywords: freezing of gait; amyloid; cholinergic; mobility; PET; imaging; MRI
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva for DNA Serum (approx. 4ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Parkinson's disease without FoG: Subjects with Parkinson's disease that do not have freezing of gait observed during motor assessment while both on or off dopaminergic medication who have undergone Brain PET imaging of 11C-DBTZ, 18F-FEOBV (vesicular acetylcholine transporter, and 11C-PIB (beta-amyloid).
  Interventions: Other: Detailed motor testing, including FoG, in PD subjects
- Parkinson's disease with FoG only while off-meds: Subjects with Parkinson's disease that have freezing of gait observed during motor assessment only while off dopaminergic medication who have undergone Brain PET imaging of 11C-DBTZ, 18F-FEOBV (vesicular acetylcholine transporter, and 11C-PIB (beta-amyloid).
  Interventions: Other: Detailed motor testing, including FoG, in PD subjects
- Parkinson's disease with FoG worse while off-meds: Subjects with Parkinson's disease that have freezing of gait observed during motor assessment while both on and off dopaminergic medication, but greater severity of FoG under off-med, who have undergone Brain PET imaging of 11C-DBTZ, 18F-FEOBV (vesicular acetylcholine transporter, and 11C-PIB (beta-amyloid).
  Interventions: Other: Detailed motor testing, including FoG, in PD subjects
- Parkinson's disease with FoG equivalent between on and off meds: Subjects with Parkinson's disease that have freezing of gait observed during motor assessment while both on and off dopaminergic medication, with no apparent effect of dopaminergic medication on FoG, who have undergone Brain PET imaging of 11C-DBTZ, 18F-FEOBV (vesicular acetylcholine transporter, and 11C-PIB (beta-amyloid).
  Interventions: Other: Detailed motor testing, including FoG, in PD subjects

INTERVENTIONS:
Other: Detailed motor testing, including FoG, in PD subjects — Subjects with PD with and without freezing of gait (FoG) will undergo a biomechanical assessment during a FoG provocation protocol in both the dopaminergic "on" and "off" state.

SUMMARY:
Early stage Parkinson disease (PD) is characterized by a 'honeymoon' phase in terms of responsiveness of motor symptoms, including gait, to dopaminergic pharmacotherapy. Advancing PD is associated with disabling axial motor complications, such as freezing of gait (FoG), with decreased or even refractory dopamine responsiveness in over 50% of patients. The management of dopamine resistant gait problems represents the most important unmet need in PD. This study will related detailed motor testing to brain PET imaging to see if certain molecules (or lack thereof) involved with neurologic transmission in the brain are involved with FoG.

DETAILED DESCRIPTION:
Early stage Parkinson disease (PD) is characterized by a 'honeymoon' phase in terms of responsiveness of motor symptoms, including gait, to dopaminergic pharmacotherapy. Advancing PD is associated with disabling axial motor complications, such as freezing of gait (FoG), with decreased or even refractory dopamine responsiveness in over 50% of patients. The management of dopamine resistant gait problems represents the most important unmet need in PD. At present, there is no biomarker of FoG in patients with PD as there is a lack of mechanistic understanding of dopamine nonresponsiveness of FoG. The investigators have previously identified cholinergic denervation as a prominent factor related to both falls and gait slowing in PD. The investigators recently identified that cortical -amyloid deposition not only associates with cognitive decline but also with postural instability and gait difficulties in PD. In this proposal, the investigators present preliminary data suggesting that FoG is associated with either cholinopathy, amyloidopathy or both in PD. The investigators propose to test the novel hypothesis that comorbid amyloidopathy may be a possible mechanistic factor underlying the poor response of FoG to dopaminergic therapy in advancing PD. In contrast, isolated cholinopathy would be expected to be associated with preserved dopamine responsiveness of FoG. For this purpose, the investigators propose to perform detailed motor, including FoG, testing in PD patients "on" and "off" their dopaminergic medications and relate this to dopaminergic 11C-dihydrotetrabenazine (DTBZ), vesicular acetylcholine transporter 18F-fluoroethoxybenzovesamicol (FEOBV) and -amyloid 11C-labeled Pittsburgh Compound-B (PIB) brain PET imaging in PD subjects with and without FoG. Furthermore, based on recent clinical observations that serotoninergic drugs, like the popular anti-depressant selective serotonin reuptake inhibitor (SSRI) drugs, are associated with significantly lower build- up of -amyloid plaques in the elderly population, and based on the investigators' subsequent observation of an intriguing inverse relationship between -amyloid plaque deposition and striatal serotoninergic terminal in PD, the investigators propose to perform an exploratory sub-study to test a new hypothesis that PD subjects with FoG will exhibit not only higher striatal -amyloid but also lower striatal serotoninergic innervation (as determined by 11C-DASB serotonin PET imaging) compared to PD subjects without FoG. If confirmed, positive findings in this study would allow the identification of different PD subgroups ('personalized medicine'), such as presence amyloidopathy or cholinopathy, to select patients for targeted pharmacotherapies to potentially prevent the development of FoG (anti-amyloid, such as serotoninergic drugs) or manage its clinical manifestation (cholinergic augmentation therapy) in order to preserve and maintain a good quality of life in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* PD based on the United Kingdom Parkinson's Disease Society Brain Bank
* Diagnostic Research Criteria with or without Freezing of Gait
* Duration of Disease > 5 years
* Mini-Mental State Examination (MMSE) > 23

Exclusion Criteria:

* Dementia
* Dementia with Lewy Bodies
* Other disorders which may resemble PD
* Subjects on neuroleptic, anticholinergic (trihexyphenidyl, benztropine) or cholinesterase inhibitor drugs
* Evidence of a stroke or mass lesion on structural brain imaging (MRI)
* Participants in whom MRI is contraindicated including, but not limited to:

  * those with a pacemaker
  * presence of metallic fragments near the eyes or spinal cord
  * cochlear implant
* Severe claustrophobia precluding MR or PET imaging
* Subjects limited by participation in research procedures involving ionizing radiation
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample recruited from the following sources
  1. UMHS Movement Disorders Clinics
  2. VA Ann Arbor HS Movement Disorders Clinic
  3. Existing studies at Functional Neuroimaging, Cognitive, and Mobility Lab at the University of Michigan
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas I Bohnen, MD PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were excluded before assignment because they showed a normal dopaminergic PET brain scan prior to motor assessment. 7 participants were excluded before assignment because they didn't consent to being recorded on camera during motor assessment. Another 7 participants were dropped for showing normal dopaminergic scan after motor assesment, which precluded them from being assigned into groups.
Period: Overall Study
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between on and Off Meds
Started | 13 | 7 | 10 | 7
Received DTBZ, PIB, and FEOVB PET Scan | 11 | 6 | 9 | 5
Completed | 11 | 6 | 9 | 5
Not Completed | 2 | 1 | 1 | 2
Not completed — Scan Limitation | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Parkinson's Disease With FoG Equivalent Between On and Off-meds: Subjects with Parkinson's disease that have freezing of gait observed during motor assessment while both on and off dopaminergic medication, with no apparent effect of dopaminergic medication on FoG, who have undergone Brain PET imaging of 11C-DBTZ, 18F-FEOBV (vesicular acetylcholine transporter, and 11C-PIB (beta-amyloid).
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds | Total
Number analyzed (Participants) | 11 | 6 | 9 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.27 (5.81) | 63.5 (8.57) | 72.78 (6.96) | 71.8 (6.94) | 68.87 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 1 | 5
  Male | 9 | 6 | 7 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 6 | 9 | 5 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 6 | 9 | 5 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 6 | 9 | 5 | 31

OUTCOME MEASURES:

1. Primary Outcome: L-DOPA Insensitivity
Description: Participants are considered as L-DOPA insensitive if their freezing of gait is not observed to be any different between motor assessment while on dopaminergic medication and off dopaminergic medication.
Time Frame: through study completion, an average of 6 months
Population: Only participants that have freezing of gait during either on or off meds motor assesment.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Freezing of Gait: L-DOPA insensitivity was assessed in a subset of participants that showed freezing of gait during either on or off medication motor examination.
Arm/Group | Participants With Freezing of Gait
Number analyzed (Participants) | 20
Participants | 5
Statistical Analysis 1: Comparison: Participants With Freezing of Gait; L-DOPA sensitivity outcome measure was modeled with 3-level hierarchical ordinal logistic regression. The null model contained only striatal DTBZ as predictor of group, the FEOVB model additionally had FEOVB tracer, and interaction model had in addition an interaction term between FEOVB and PIB tracer. Model comparisons were performed using Chi-Square goodness of fit test; Test type: Other; p = 0.00468, ChiSq Goodness of Fit Test — The p-value is derived from model comparison between the FEOVB model and the FEOVB*PIB interaction model; Standardized β Coefficient = -2.256

2. Primary Outcome: Striatal FEOVB PET Binding
Description: Parametric distribution volume ratio (DVR) of FEOVB, a cholinergic PET tracer, in the striatum.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: distribution volume ratio
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds
Number analyzed (Participants) | 11 | 6 | 9 | 5
distribution volume ratio | 4.89 (0.7) | 5.01 (0.69) | 4.30 (0.81) | 4.06 (0.80)

3. Primary Outcome: Striatal DTBZ PET Binding
Description: Parametric distribution volume ratio (DVR) of DTBZ, a dopaminergic PET tracer, in the striatum.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: distribution volume ratio
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds
Number analyzed (Participants) | 11 | 6 | 9 | 5
distribution volume ratio | 1.93 (0.36) | 1.76 (0.24) | 1.59 (0.20) | 1.76 (0.35)

4. Primary Outcome: Striatal PIB PET Binding
Description: Parametric distribution volume ratio (DVR) of PIB, an amyloid PET tracer, in the striatum.
Time Frame: through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: distribution volume ratio
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds
Number analyzed (Participants) | 11 | 6 | 9 | 5
distribution volume ratio | 1.08 (0.11) | 1.15 (0.08) | 1.12 (0.12) | 1.02 (0.07)

5. Secondary Outcome: Serotonergic Innervation of Striatum and Freezing
Description: Serotonergic innervation of striatum as assessed by DASB PET scan across freezer groups.
Time Frame: through study completion, an average of 6 months
Population: Limited subset of participants that underwent a serotonergic DASB PET scan.
Measure: Number; unit: Parametric DVR
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds
Number analyzed (Participants) | 1 | 0 | 1 | 1
Parametric DVR | 1.741856 |  | 1.120202 | 1.796165

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Arm/Group | Parkinson's Disease Without FoG | Parkinson's Disease With FoG Only While Off-meds | Parkinson's Disease With FoG Worse While Off-meds | Parkinson's Disease With FoG Equivalent Between On and Off-meds
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7 | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7 | 0/10 | 0/7

LIMITATIONS AND CAVEATS:
The sample was predominantly male limiting generalization to the broader PD patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03647137/Prot_SAP_ICF_000.pdf